CLINICAL TRIAL: NCT05992883
Title: NSAID Injection Versus Corticosteroid Injection for Basilar Thumb Arthritis: A Randomized, Controlled Trial
Brief Title: NSAID Injection Versus Corticosteroid Injection for Basilar Thumb Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marco Rizzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-005275
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Thumb Osteoarthritis
Keywords: Injection; Steroid; NSAID; Thumb Arthritis; CMC Arthritis
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Triamcinolone

STUDY DESIGN:
Intervention Model Description: This trial will be a single center, comparative, randomized (1:1 ratio), prospective, double-blind trial with two groups evaluated concurrently. One group will be given triamcinolone injections while the second, experimental group will receive ketorolac injections.
Who Masked: Participant, Care Provider
Masking Description: After enrollment and completion of the initial clinical evaluation, patients will undergo the injection procedure while blinded to the medication they receive. The injecting physician will also be blinded to the medication being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non-steroidal anti-inflammatory drug (NSAID) (Experimental): Patients will proceed to their injection appointment within 4 weeks of their initial evaluation. At the injection appointment, patients will receive an injection containing 1.0 mL of ketorolac 15 mg/mL (15 mg total of ketorolac).
  Interventions: Drug: Ketorolac
- Corticosteroid (Active Comparator): Patients will proceed to their injection appointment within 4 weeks of their initial evaluation. At the injection appointment, patients will receive an injection containing 0.5 mL of triamcinolone 40 mg/mL (20 mg total of triamcinolone).
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Ketorolac — Intervention will be an injection containing 1.0 mL of ketorolac 15 mg/mL (15 mg total of ketorolac).
  Other Names: Toradol
  Arms: Non-steroidal anti-inflammatory drug (NSAID)
Drug: Triamcinolone — Intervention will be an injection containing 0.5 mL of triamcinolone 40 mg/mL (20 mg total of triamcinolone).
  Arms: Corticosteroid

SUMMARY:
The Researchers are trying to compare two different types of intraarticular injections (injection in the joint) for treating the symptoms of moderate to advanced basilar thumb arthritis. One injection is ketorolac (an NSAID) and the other is triamcinolone (a corticosteroid).

DETAILED DESCRIPTION:
Cartilage degeneration resulting in osteoarthritis is the most common and costly musculoskeletal disorder in the United States, with basilar thumb arthritis being one of the most common manifestations of this disease. Despite its prevalence and previous research on treatments for the disease, there is a dearth of efficacious and low-cost interventions for trapeziometacarpal arthritis. Of these nonoperative interventions, intraarticular corticosteroid injections are the most popular and have the most evidence indicating their benefit. However, long-term use of corticosteroids has a well-established degenerative effect that is counterproductive to preserving cartilage and bone of the CMC joint. Novel, disease-modifying osteoarthritis treatments such as platelet rich plasma and human recombinant bone morphogenic protein 7, among others, are alternative options for patients. Many of these are currently in advanced development, but to date none have achieved FDA approval, and all are significantly more expensive and have limited availability compared to intraarticular corticosteroids.

Although used infrequently, non-steroidal anti-inflammatory drugs (NSAIDs) are another modality of nonoperative intervention for basilar thumb arthritis. Intraarticular injections of NSAIDs have demonstrated success in alleviating the symptoms of primary arthritis in the hip and knee without concern of systemic side effects compared to oral NSAID use. Additionally, injectable NSAIDs are significantly more cost-effective compared to other injectables and do not have the chondrotoxic profile of corticosteroids. However, there are few studies directly comparing intraarticular NSAID use to other injectable therapies.

Given the potential clinical and economic benefits of injectable NSAID therapy, we propose a clinical trial investigation examining the efficacy of intraarticular ketorolac versus intraarticular triamcinolone in treating symptoms of moderate to advanced primary osteoarthritis of the basilar thumb. The prospect of successfully alleviating symptoms of joint degeneration without propagating the progression of disease would be invaluable to the thousands of patients in the Mayo Clinic system and elsewhere afflicted with basilar thumb arthritis without the means or ability to pursue stem cell therapeutics or more definitive, operative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults >40 years of age
* Pain at the thumb base brought on by direct pressure (grind test) and with movement
* Pain resistant to previous conservative management (including over the counter medications (ibuprofen/acetaminophen), icing, splinting/braces, or topical analgesics)
* Radiological observation indicative of arthritis based on the Eaton-Littler classification system (stages 1 through 4)
* Patient understands the protocol and signed the informed consent
* Patient is covered by health insurance

Exclusion Criteria:

* • Known allergy to either of the treatment products
* Patient's analgesic treatment regimen or other modalities of managing symptoms/pain associated with their hand pathology was modified within four weeks before trial inclusion
* Symptomatic Scaphoid-trapezial arthritis present
* Localized or systemic infection
* Previous thumb surgery on study thumb
* Previous thumb injury on study thumb
* Patient with inflammatory arthritis (e.g., rheumatoid arthritis, psoriatic arthritis)
* Severe and/or uncontrolled hypertension
* De Quervain tendinopathy present
* History of injection to the trapeziometacarpal joint on study thumb within the previous 6 weeks
* Uncontrolled diabetes
* Pregnant or lactating females. Female participants of childbearing potential must have a negative pregnancy test before the injection. Women without childbearing potential (ie., surgically sterile with hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy OR ≥ 12 months of amenorrhea and at least 50 years of age) are eligible to participate without completing a pregnancy test.
* Immunodeficient patients
* Patients that are currently using nicotine products, or who have quit in the last 12 months
* Patients under guardianship, curatorship, or are otherwise not self-sufficient
* Patients participating in another clinical research trial which interferes with this study protocol or outcomes
* Patients unable to follow the protocol in the investigators' judgement.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of Pain | At initial evaluation and then 1 month, 3 months, 6 months, and 1 year post-injection.
  Patient-reported VAS score with both motion and rest of the CMC joint. The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 = no pain to 10 = worst pain. Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.

SECONDARY OUTCOMES:
Michigan Hand Outcomes Questionnaire (MHQ) | At initial evaluation and then 1 month, 3 months, 6 months, and 1 year post-injection.
  The Michigan Hand Outcomes Questionnaire (MHQ) is patient-reported. An overall MHQ score can be obtained by summing the scores for all six scales after reversing the pain scale (pain=100-pain score) and then dividing by six. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance.
Grip Strength | At initial evaluation and then 1 month, 3 months, 6 months, and 1 year post-injection.
  Grip strength measured with a dynamometer, reported in kilograms. Measurements will be performed three times, with the mean value of the three repetitions used as the reported value.
Apposition Strength | At initial evaluation and then 1 month, 3 months, 6 months, and 1 year post-injection.
  Apposition strength measured with a dynamometer, reported in kilograms. Measurements will be performed three times, with the mean value of the three repetitions used as the reported value.
Opposition Strength | At initial evaluation and then 1 month, 3 months, 6 months, and 1 year post-injection.
  Opposition strength measured with a dynamometer, reported in kilograms. Measurements will be performed three times, with the mean value of the three repetitions used as the reported value.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Rizzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials